CLINICAL TRIAL: NCT05479708
Title: Postoperative ctDNA-based Minimal Residual Disease Detection for Resected Pancreatic Adenocarcinoma: A Prospective Observational Cohort Study
Brief Title: ctDNA-based Minimal Residual Disease Detection for Resected Pancreatic Adenocarcinoma
Status: Enrolling by invitation | Type: Observational
Sponsor: BAIYONG SHEN (Other)
Collaborators: GeneCast Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, BAIYONG SHEN, Professor, Ruijin Hospital
Organization: Ruijin Hospital (Other)
Other Study IDs: D-P220426-MRD-RJ-1
Record Dates: First submitted 2022-07-28; First posted 2022-07-29 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Pancreatic Cancer Resectable
Keywords: circulating tumor DNA; minimal residual disease
MeSH Terms: conditions — Neoplasm, Residual

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Matched tumor tissues, plasma samples and blood cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: ctDNA-based MRD detection — Postoperative circulating tumor DNA (ctDNA)-based minimal residual disease (MRD) detection for predicting relapse and survival benefit

SUMMARY:
Short-term relapse and poor survival are prevalent in patients with pancreatic adenocarcinoma (PAAD) after surgeries. Despite the importance of adjuvant treatments for resected PAAD patients, there is currently no suitable biomarker to identify those individuals with high risk of recurrence and inform therapeutic decision making. In this study, we aim to examine whether postoperative circulating tumor DNA (ctDNA) could be used as a biomarker for early detection of minimal residual disease (MRD) and predicting relapse in resected PAAD through high-depth targeted next-generation sequencing.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically diagnosed pancreatic adenocarcinoma (stage I-III)
* KRAS mutations identified in resected tumor tissues
* Margin negative (R0) or no imaging recurrence/metastasis and CA 19-9<37 U/ml in postoperative 4-8 weeks (before adjuvant chemotherapy)
* Receiving adjuvant chemotherapy
* ECOG 0-2
* Signed informed consent

Exclusion Criteria:

* With serious internal medicine diseases, infectious diseases, other solid tumors (except PAAD) or hematologic disorders
* Distant organ metastasis or malignant ascites
* Receiving neo-adjuvant therapy before surgery
* Imaging recurrence/metastasis or CA 19-9>37 U/ml in postoperative 4-8 weeks (before adjuvant chemotherapy)
* Pregnant or breastfeeding at time of enrollment
* Prior transplantation of bone marrow, stem cell or organ

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The pathologically diagnosed stage I-III PAAD patients who underwent resections carried KRAS mutations in tumor tissues. Margin negative (R0) or no imaging recurrence/metastasis and CA 19-9<37 U/ml in postoperative 4-8 weeks (before adjuvant chemotherapy).
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-08-09 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Death and overall survival | 3 years
  Overall survival difference between MRD-positive and MRD-negative patients

CONTACTS AND LOCATIONS:
Overall Officials: Baiyong Shen, Ph.D, Principal Investigator — Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine
Locations (1):
- Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No